CLINICAL TRIAL: NCT04156698
Title: A Phase II, Single-center, Open-label, Single-arm Study of Induction Chemotherapy Combined With Immunotherapy for Locally Advanced Hypopharyngeal Carcinoma
Brief Title: Induction Chemotherapy Combined With Immunotherapy for Locally Advanced Hypopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: zhouliang
Record Dates: First submitted 2019-11-06; First posted 2019-11-07 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Hypopharyngeal Carcinoma; Immunotherapy; Chemotherapy
Keywords: Locally advanced hypopharyngeal squamous cell carcinoma; Programmed death protein - 1 inhibitor; Camrelizumab; Objective response rate; Safety profiles
MeSH Terms: conditions — Hypopharyngeal Neoplasms | interventions — Docetaxel; Home Environment; Cisplatin; Capecitabine; camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab (PD-1 inhibitor) group (Experimental): Induction chemotherapy combined with immunotherapy (TPF + Camrelizumab), q3w, 3 cycles in total:
  Docetaxel (domestic) 75 mg/m2 i.v. d1, Cisplatin 25 mg/m2 i.v. d1-3, Capecitabine 800 mg/m2 po bid d1-d14, Camrelizumab 200mg i.v. d1;
  Radical radiotherapy plus concurrent immunotherapy (CR or PR):
  Radiotherapy: Using intensity-modulated radiation therapy (IMRT). Primary site: GTV dose 66 (2.2Gy / fraction)-70 Gy (2Gy / fraction)；CTV 1.6-1.9 Gy / fraction. Cervical lymph nodes: Radiotherapy plan is the same as the radiotherapy plan of original site; Concurrent immunotherapy : Camrelizumab 200mg i.v. d1, d22;
  Maintenance period:
  After completing concurrent chemoradiotherapy combined with immunotherapy, Camrelizumab 200 mg q3w will be given up to 12 months (calculated from the time of the first dose of PD-1 immunotherapy).
  Interventions: Drug: Docetaxel; Drug: Cisplatin; Drug: Capecitabine; Drug: Camrelizumab

INTERVENTIONS:
Drug: Docetaxel — Docetaxel is a chemotherapy drug.
  Other Names: Docetaxel (domestic)
Drug: Cisplatin — Cisplatin is a chemotherapy drug.
  Other Names: chemotherapy drug
Drug: Capecitabine — Capecitabine is a chemotherapy drug.
  Other Names: chemotherapy drug
Drug: Camrelizumab — Camrelizumab is a humanized anti-PD1 IgG4 monoclonal antibody.
  Other Names: Anti-PD-1 Antibody (Jiangsu Hengrui)

SUMMARY:
This is a single-center, multidisciplinary, open-label, single-arm prospective clinical study.

DETAILED DESCRIPTION:
In this study, 51 patients with hypohparyngeal carcinoma will be enrolled, These patients who have locally advanced-stage disease, including TNM stage cT3-4aN0-2M0 (AJCC 7th) and require a total laryngectomy as an initial therapy. Patients who achieved a CR or PR at the primary site after three cycles of TPF-regimen chemotherapy combined with immuotherapy will be referred for definitive RT and immuotherapy, while patients who received an evaluation of PD or SD at the primary site were referred for surgery followed by adjuvant RT/CRT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have histologically confirmed hypopharyngeal squamous cell carcinoma and require total laryngectomy, including the piriform fossa, postcricoid region, and posterior pharyngeal wall with TNM stage cT3-4aN0-2M0(AJCC 7th).
2. Able to understand and willing to sign a written informed consent document.
3. Age≥ 18 and≤ 70 years.
4. Male or female.
5. Performance status of ECOG 0-2.
6. Expected lifetime > 6 months.
7. Normal blood test, hepatic and renal functions. Normal hearing. Blood test: WBC≥4.0×109/L，ANC≥2.0×109/L，PLT≥100×109/L，HGB≥100g/L；Hepatic function: ALT、AST< upper limit of normal. Kidney function: Serum creatinine < upper limit of normal value, and creatinine clearance rate ≥ 60 ml/min（Cockcroft-Gault formula）. Cardiac ultrasonography left ventricular ejection fraction >50%.
8. No prior allergic reaction to biological agents and/or ingredient in the drug.
9. No drug abuse.
10. Good compliance.
11. No other important related diseases (such as other tumors, severe heart, lung and central nervous system diseases, etc.).
12. Negative pregnancy test (for female patients with fertility).
13. Male patients with fertility and female patients with fertility and pregnancy risk must agree to use contraceptive methods throughout the study period, and continued until at least 6 months after the last dose of cisplatin and 30 days after the last dose of PD-1 antibody/placebo (whichever occurs later). Female patients who do not have fertility (ie meet at least one of the following criteria): Have undergone hysterectomy and/or bilateral oophorectomy with archival records, medically confirmed ovarian function decline; In postmenopausal state. It is defined as: At least 12 months of continuous menstruation without other pathological or physiological reasons, and the status confirmed by serum follicle stimulating hormone (FSH) levels is consistent with postmenopausal status.

Exclusion Criteria:

1. Patients with cervical lymph node cN3.
2. Have a history of other cancers in the past five years, radical or untreated prostate cancer (Gleason score ≤ 6), or complete treatment of breast ductal carcinoma in situ, except for patients with cured skin basal cell carcinoma or squamous cell skin cancer.
3. Patients with target lesions who have received radiation therapy or surgery (except biopsy).
4. Patients who have previously used chemotherapy, immunotherapy, or biological targeted therapy for primary tumors
5. Patients who have participated in other clinical trials within 4 weeks before the test.
6. Any of the following conditions in the first 6 months of random grouping: myocardial infarction, severe/unstable angina, coronary artery/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, patients with transient ischemic attack or symptomatic pulmonary embolism.
7. Patients with hypertension who cannot control well through single antihypertensive medication (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg);
8. Patients with grade I or above coronary heart disease, arrhythmia (including men with a QTc interval >450 ms, women >470 ms), and cardiac insufficiency.
9. Urinary protein was greater than ++ and 24-hour urinary protein quantification >1.0 g.
10. Many factors that affect oral medications (such as inability to swallow, nausea, vomiting, chronic diarrhea, and intestinal obstruction).
11. Patients with abnormal coagulation function（INR>1.5、APTT>1.5 ULN）and bleeding tendency.
12. Patients with a history of psychotropic substance abuse that is active or has a mental disorder.
13. Patients who required systemic treatment with corticosteroids (>10 mg prednisone equivalent daily) or other immunosuppressive agents within 2 weeks prior to the first use of the study drug.
14. Patients with a history of severe allergies or allergies; patients with active autoimmune diseases that may worsen when receiving immunostimulants; patients with type 1 diabetes, vitiligo, psoriasis, or hypothyroidism or hyperthyroidism who do not require immunosuppressive therapy are eligible to participate in the study.
15. Patients who have previously been diagnosed with immunodeficiency or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related diseases. Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (HBV) surface antigen is positive at screening, or patients with positive HCV RNA [ribonucleic acid] when positive for anti-HCV antibody screening test.
16. Vaccination within 4 weeks prior to randomization, except for inactivated vaccines.
17. Pregnant or lactating women who are in the reproductive period but have not taken effective contraceptive measures.
18. The investigator believes that it is inappropriate for individuals to participate in the trial: having, for example, severe acute or chronic medical conditions (including immune colitis, inflammatory bowel disease, non-infectious pneumonia, pulmonary fibrosis) or mental illness (including recent time [within the past year] or active suicidal ideation or behavior) .
19. With a history of tuberculosis or antituberculosis treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2023-04-16 (Actual); Study Completion 2026-01-16 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 9 weeks
  The proportion of patients with partial and complete response as defined by RECIST 1.1 after induction therapy

SECONDARY OUTCOMES:
LPR | 3 years
  Larynx preservation rate
PFS | 3 years
  Progression free survival
MFS | 3 years
  Metastasis free survival
OS | 3 years
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Liang Zhou, PhD., Principal Investigator — Eye & ENT Hospital, Fudan University
Locations (1):
- Eye & ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China